CLINICAL TRIAL: NCT05048979
Title: Telehealth to Improve Functional Status and Quality of Life in Veterans With PAD (CDA 20-073)
Brief Title: Telehealth to Improve Functional Status and Quality of Life in Veterans With PAD
Acronym: MOVE-IT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDX 21-006
Record Dates: First submitted 2021-09-01; First posted 2021-09-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Enrollment in a 12-week, 3 day a week, aerobic training program in a self-selected location. The exercise training will be via telehealth. Arm 1 will receive aforementioned intervention. Arm 2 will received no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): Prospective pre-post pilot study design. (N=54)
  Interventions: Other: Exercise
- No exercise (No Intervention): Prospective cohort study design. (N=100)

INTERVENTIONS:
Other: Exercise — Telehealth-facilitated supervised exercise program. Veterans with PAD will be enrolled in a 12-week, 3 day a week, aerobic training program in a self-selected location.
  Arms: Exercise

SUMMARY:
The present study aims to increase Veteran access to supervised exercise therapy and expand its role in improving functional status, quality of life, and cardiovascular risk profile of Veterans with PAD.

DETAILED DESCRIPTION:
The investigators will use the VA Telehealth service to deploy a remotely accessible supervised exercise training program and evaluate whether a telehealth-based intervention can improve walking performance, quality of life, and ultimately cardiac risk in Veterans with PAD. The impetus for the current proposal stems from the following: 1) over 50% of VA-enrolled Veterans live in rural communities; 2) Veterans with PAD are older (mean age, 70 years), further increasing their risk for functional decline; and 3) there is a significant lack of access to facility-based supervised exercise training for Veterans with PAD. The objectives include the following:

1. To develop a telehealth-facilitated exercise intervention for Veterans with PAD that serves as a Veteran centric new model of care.
2. To integrate Veteran preferences into the development of a telehealth-facilitated supervised exercise program.
3. To assess the long-term patterns of functional impairment and quality of life among Veterans with PAD not undergoing supervised exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAD, defined as a history of an ankle-brachial index (ABI) of 0.90, prior revascularization of a lower limb for symptomatic disease more than 30 days prior to presentation, or ABI >0.90 with evidence of PAD based on noninvasive vascular laboratory testing or angiography

  * [and presence of claudication, defined as fatigue, discomfort, cramping or pain of vascular origin in the muscles of the lower extremities that is consistently induced by exercise and consistently relieved by rest within 10 minutes.]
* In addition, participants will require access to cellular signal at place of residence and/or exercise location

Exclusion Criteria:

* Justification for exclusion criteria centers on inability to safely participate in the remote intervention. Specific exclusion criteria includes the following:
* major lower extremity amputation
* critical limb ischemia
* inability to ambulate without a walker or wheelchair
* significant visual or hearing impairment
* individuals whose function is limited by severe conditions such as severe ischemic heart disease or > Class II NYHA heart failure
* individuals capable of ambulating at a level comparable to the amount of exercise to be prescribed at baseline
* individuals currently enrolled in another exercise trial or cardiac rehab program
* individuals with uncontrolled psychiatric illness or dementia
* categorically vulnerable

  * pregnant women, prisoners, children, or persons who lack decision-making capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | At 3-months
  Participants will be asked to walk in an unobstructed 100-ft hall for 6 continuous minutes with the goal of walking the greatest distance possible. Participants are allowed to stop and rest (standing or sitting), but the stopwatch will continue to run. The key outcome is distance walked. This outcome will be evaluated at the 3-month mark.
Walking impairment Questionnaire (WIQ) | At 3-months
  Will evaluate the following: 1) symptoms while walking (typical and atypical); 2) perceived difficulty walking defined distances (ranging from walking indoors to 1,500 feet or 5 blocks); 3) and perceived difficulty walking defined speeds; and 4) ability to climb stairs. Assessments are made on a graded scale from 0 to 4. A difficulty score a 0 represents very difficult and 4 represents no difficulty. The graded scores are multiplied by prespecified weights for each distance, speed, or number of flights of stairs. The products are then summed and divided by the maximum possible score ranging from 0 (inability to perform the task) to 100 (no difficulty performing the task). This outcome will be evaluated at the 3-month mark.
Vascular quality of life questionnaire (VascuQol) | At 3-months
  The Vascular Quality of Life Questionnaire (VascuQol) is a PAD specific and commonly used health related quality of life questionnaire with positive responsiveness correlated to both clinical improvement and deterioration on short and long term follow-up subsequent to treatment interventions. The VascuQol consists of items that span five domains (pain, symptoms, activities, emotional, and social). Each item is scored on a seven-point rating scale, where 1 represents the worst and 7 the best possible score. A sum score is calculated by dividing the sum all items by 25. This outcome will be evaluated at the 3-month mark.
Flourish measure | At 3-months
  The Flourish Measure is a composite evaluation of human well-being with excellent viability, and applicability in both community and workplace. The Flourish Measure consists of 12 questions that span 6 domains (happiness and life satisfaction, mental and physical health, meaning and purpose, character and virtue, close social relationships, financial and material stability). Each item is scored on an eleven-point rating scale of 0-10 with higher scores indicating favorable responses. Scores are calculated by summing the scores of all six domains. This outcome will be evaluated at the 3-month mark.
Claudication onset time | At 3-months
  The walking time at which the subjects first experienced lower extremity pain. This outcome will be evaluated at the 3-month mark.
Peak walking time | At 3-months
  Walking time at which ambulation cannot continue due to maximal lower extremity pain. This outcome will be evaluated at the 3-month mark.
10 meter walk | At 3-months
  Time it takes subject to walk 10 meters. Measured in seconds. This outcome will be evaluated at the 3-month mark.
Balance test | At 3-months
  Subject balance evaluated by having them stand with feet side-by-side, semi-tandem, and then tandem. For each stance outcome is measures as yes or no. This outcome will be evaluated at the 3-month mark.
30-sec arm curls | At 3-months
  Measured in number of repetitions (8 pound weight for men and 5 pound weight for women). This outcome will be evaluated at the 3-month mark.
30-sec-chair stands | At 3-months
  Measured in number of repetitions. This outcome will be evaluated at the 3-month mark.
8 feet get up and go walk | At 3-months.
  Time it takes to go from sitting to standing and walking 8 feet. Measured in seconds. This outcome will be evaluated at the 3-month mark.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Antonio Gutierrez, MD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No